CLINICAL TRIAL: NCT06020976
Title: Pattern of Autoimmune Hepatitis in Children In Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fathy Mohamed Abdelhakam, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-23-07-10MS
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liver biobsy — all pationt will be subjected yo liver biobsy to confirm diagnosis

SUMMARY:
Autoimmune hepatitis (AIH) is a progressive inflammatory liver disorder of unknown etiology. If left untreated, it progresses to liver cirrhosis and liver failure.

Diagnosis of AIH relies on the exclusion of other causes of liver disease and the presence of positive clinical, biochemical, and histological criteria.

AIH has a very wide spectrum of clinical presentations ranging from being asymptomatic to an acute severe fulminant disease.

It may be associated with other autoimmune disorders such as thyroiditis, type 1 diabetes, vitiligo, inflammatory bowel disease, or juvenile idiopathic arthritis.

Biochemical features of AIH include elevation of serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), and immunoglobulin G (IgG) in addition to autoantibodies.

Liver biopsy is recommended in any patient with suspected autoimmune hepatitis where interface hepatitis is the hallmark of the disease.

Immunosuppression is the mainstay of therapy in AIH. Prednisone is administered as the initial therapy either alone or in combination with azathioprine.

Liver transplantation is indicated in patients who develop fulminant hepatic failure that is unresponsive to corticosteroids and in patients who develop end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: under 18 years old.
* Both sex.
* children suffering from manifestations of Autoimmune Hepatitis. Children previously Diagnosed with Autoimmune Hepatitis

Exclusion Criteria:

* Patient infected with hepatitis B or C.
* Patient had autoimmune hepatitis after liver transplantation.
* Patients not respond to steroids and immunosuppressive therapy. Other Causes of acute and chronich hepatitis like wilson disease and Metabolic liver Diseases

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Age: under 18 years old.
  * Both sex.
  * children suffering from manifestations of Autoimmune Hepatitis. Children previously Diagnosed with Autoimmune Hepatitis-
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
liver biobsy | 1 year
  to confirm charachterstic features of autoimmune hepatitis in liver biobsy as interface hepatitis portal inflammation
autoantibody | 1 year
  Autoantibodies will be considered positive and clinically significant when present at a dilution ≥1:20 for antinuclear antibody (ANA) and smooth muscle antibody (SMA) or ≥1:10 for liver kidney microsomal (anti-LKM-1).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mieli-Vergani G, Heller S, Jara P, Vergani D, Chang MH, Fujisawa T, Gonzalez-Peralta RP, Kelly D, Mohan N, Shah U, Murray KF. Autoimmune hepatitis. J Pediatr Gastroenterol Nutr. 2009 Aug;49(2):158-64. doi: 10.1097/MPG.0b013e3181a1c265. PMID 19561543
- [Background] Maggiore G, Nastasio S, Sciveres M. Juvenile autoimmune hepatitis: Spectrum of the disease. World J Hepatol. 2014 Jul 27;6(7):464-76. doi: 10.4254/wjh.v6.i7.464. PMID 25067998
- [Background] Manns MP, Czaja AJ, Gorham JD, Krawitt EL, Mieli-Vergani G, Vergani D, Vierling JM; American Association for the Study of Liver Diseases. Diagnosis and management of autoimmune hepatitis. Hepatology. 2010 Jun;51(6):2193-213. doi: 10.1002/hep.23584. No abstract available. PMID 20513004
- [Background] Mieli-Vergani G, Vergani D, Czaja AJ, Manns MP, Krawitt EL, Vierling JM, Lohse AW, Montano-Loza AJ. Autoimmune hepatitis. Nat Rev Dis Primers. 2018 Apr 12;4:18017. doi: 10.1038/nrdp.2018.17. PMID 29644994